CLINICAL TRIAL: NCT03838822
Title: Kinetics of Metabolic Cofactors After Oral Supplementation in Healthy Subjects
Brief Title: Kinetics of Metabolic Cofactors in NAFLD
Acronym: NAFLDCOFCAL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Chalmers University of Technology (Other)
Responsible Party: Principal Investigator, Hanns-Ulrich Marschall, Professor, University Hospital Consultant, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cofactor Calibration 1.0
Record Dates: First submitted 2019-02-04; First posted 2019-02-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: nicotinamid riboside; L-carnitine; L-serine; N-acetylcystein
MeSH Terms: interventions — 5,11-methenyltetrahydrohomofolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Oral administration of cofactors, 1g nicotinamide riboside, 3g L-carnitine, 20g serine and 5g N-acetylcystein, first as single compounds, then combined, on 5 days
  Interventions: Dietary Supplement: Cofactors

INTERVENTIONS:
Dietary Supplement: Cofactors — Oral administration of 1g nicotinamide riboside, 3g L-carnitine, 20g serine and 5g N-acetylcystein, first as single compounds, then combined, on 5 days

SUMMARY:
There is a strong correlation between major adverse health consequences of obesity and development of non-alcoholic fatty liver disease (NAFLD). NAFLD is characterized by abnormal hepatic accumulation of triglycerides and other lipids. It has become a worldwide health problem that accelerates cirrhosis, type 2 diabetes mellitus (T2DM), and especially premature cardiovascular morbidity and mortality.

The plasma level of glutathione (GSH) is typically depleted in individuals with metabolism related disorders. However, cellular GSH levels cannot be increased by supplementing GSH and it must be synthesized within the liver either de novo or by salvation pathway. The level of GSH is not enough to maintain and regulate the thiol redox status of the liver in subjects with high hepatic steatosis at fasting stage due to the depletion of glycine. Glycine can be synthesized via the interconversion of serine. It has been shown that the serine synthesis is downregulated in patients with NAFLD and supplementation of serine has attenuated alcoholic fatty liver by enhancing homocysteine metabolism in mice and rats. Depleted liver glutathione is also restored by the administration of N-acetylcystein as in acetaminophen poising. L-carnitine and nicotinamide that both stimulate the transfer of fatty acids from cytosol to mitochondria have been identified as two additional cofactors that are depleted in patients with NAFLD.

In this study, the kinetics in blood of pivotal metabolic cofactors, serine, L-carnitine, N-acetylcystein and nicotinamide after single and simultaneous dietary supplementation, are measured.

DETAILED DESCRIPTION:
In 10 healthy subjects with BMI <30 kg/m2 the plasma concentrations of 4 natural compounds (nicotinamide riboside, L-carnitine, L-serine and N-acetylcystein) are measured by ultra-performance liquid chromatography-tandem mass spectrometry (UPLCMSMS) after individual and combined administration, on five consecutive days and at every hour during 9 hours after administration. The study will start at 8:00 every morning and at each time point, blood samples will be collected.

The taste and any potential sensing of the co-factors such as vertigo, nausea, bowel movement will be recorded.

Each participant will receive one oral dose of Day 1: 1 g nicotinamide riboside; Day 2: 3 g L-carnitine; Day 3: 5 g N-acetylcystein; Day 4: 20 g L-serine; Day 5: combined 1 g nicotinamide riboside, 3 g L-carnitine, 5 g N-acetylcystein, and 20 g L-serine

In addition, untargeted metabolomics analysis as well as O-link proteomics analysis we be performed to study effect of the administered cofactors.

ELIGIBILITY:
Inclusion Criteria:

Healthy without any medication, no smokers, no obesity

Exclusion Criteria:

Any known disease, obesity

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Changes of plasma levels of nicotinamide riboside measured by mass spectrometry | Twenty-four hours after administration
  Plasma levels of nicotinamide riboside by UPLCMSMS at 8 time points during 24h after administration
Changes of plasma levels of L-carnitine measured by mass spectrometry | Twenty-four hours after administration
  Plasma levels of L-carnitine (nM) measured by UPLCMSMS at 8 time points during 24h after administration
Changes of plasma levels of L-serine measured by mass spectrometry | Twenty-four hours after administration
  Plasma levels of L-serine (nM) measured by UPLCMSMS at 8 times points during 24h after administration
Changes of plasma levels of N-acetylcystein measured by mass spectrometry | Twenty-four hours after administration
  Plasma levels of N-acetylcystein (nM) measured by UPLCMSMS at 8 times points during 24h after administration

SECONDARY OUTCOMES:
Changes in the plasma level of metabolites associated with the supplementation of metabolic co-factors. | Twenty-four hours after administration of combined cofactors
  Untargeted metabolomic analysis using mass spectrometry. (Untargeted = not pre-specified in terms of outcome)
Changes in the plasma level of inflammation-related proteins associated with the supplementation of metabolic co-factors. | Twenty-four hours after administration of combined cofactors
  Changes in the plasma level of inflammation related proteins associated with the supplementation of metabolic co-factors.

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Ulrich Marschall, Prof, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Hanns-Ulrich Marschall, Gothenburg
  - Sahlgrenska Academy, Gothenburg

IPD SHARING:
Plan to Share IPD: No